CLINICAL TRIAL: NCT03764046
Title: Development and Validation of New "SNU Illustrated Pain Rating Scale" for Effective Assessment of Acute Postoperative Pain: a Comparative Study With Numeric Rating Scale
Brief Title: Development and Validation of New "SNU Illustrated Pain Rating Scale" as a Tool for Postoperative Pain Assessment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Other Study IDs: SNUMR2-2
Record Dates: First submitted 2018-11-30; First posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Pain Measurement; Acute Pain; Postoperative Pain; Anesthesia; Surgery
Keywords: Pain Measurement; Acute Postoperative Pain
MeSH Terms: conditions — Acute Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The numeric rating scale (NRS), one of the most widely used pain scales in clinical practice, although convenient, is often subject to bias because it requires abstract thinking from both the patient and the evaluator. Compared to numbers, traumatic pain, when visualized appropriately, has potential advantage as a means to indicate and communicate the severity of pain. Given that they are standardized in terms of body parts, wound size, and bleeding volume, illustrations of traumatic pain along with external somatic stimuli that caused it can be used to serve as effective visual anchors to supplement a pain scale by giving more concrete information to the patient. The purpose of this study is to develop Seoul National University Illustrated Pain Scale(SNUIPS) using pictures of traumatic pain, and verify the validity and effectiveness of this scale in comparison with those of NRS.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing a gynecological or orthopedic surgery under general anesthesia
* Administered with intravenous patient-controlled analgesia for postoperative pain control
* American Society of Anesthesiologists physical status class I-III patients

Exclusion Criteria:

* Contraindicated against fentanyl
* Unable to communicate
* Aged less than 18, or more than 79
* Weighs less than 40kg or more than 89kg
* Has severe heart disease(s)
* Pregnant

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 adult patients undergoing postoperative pain control after a gynecological or orthopedic surgery at Seoul National University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Scores (NRS) | 24 hours after surgery
  Self-reported pain intensity based on numeric rating scale evaluated after 24 hours after surgery. Each item is scored from 0 to 10 (0 = no pain; 10 = worst imaginable pain). Retrospective assessment of peak postoperative pain intensity will be included in addition to evaluation of current pain intensity.
Postoperative Pain Scores (NRS) | 24.5 hours after surgery
  Self-reported pain intensity based on numeric rating scale evaluated after 24.5 hours after surgery for validation in terms of test-retest reliability of the scale. Each item is scored from 0 to 10 (0 = no pain; 10 = worst imaginable pain). Retrospective assessment of peak postoperative pain intensity will be included in addition to evaluation of current pain intensity.
Postoperative Pain Scores (NRS) | 48 hours after surgery
  Self-reported pain intensity based on numeric rating scale evaluated after 48 hours after surgery for assessment of sensitivity to change. Each item is scored from 0 to 10 (0 = no pain; 10 = worst imaginable pain).
Postoperative Pain Scores (SNUIPS) | 24 hours after surgery
  Self-reported pain intensity based on Seoul National University Illustrated Pain Scale evaluated after 24 hours after surgery. Each item is scored using illustrations that corresponds to 0-10 levels of traumatic pain, beginning from 'no injury and/or pain' to 'causalgia'. Retrospective assessment of peak postoperative pain intensity will be included in addition to evaluation of current pain intensity.
Postoperative Pain Scores (SNUIPS) | 24.5 hours after surgery
  Self-reported pain intensity based on Seoul National University Illustrated Pain Scale evaluated after 24.5 hours after surgery. Each item is scored using illustrations that corresponds to 0-10 levels of traumatic pain, beginning from 'no injury and/or pain' to 'causalgia'. Retrospective assessment of peak postoperative pain intensity will be included in addition to evaluation of current pain intensity.
Postoperative Pain Scores (SNUIPS) | 48 hours after surgery
  Self-reported pain intensity based on Seoul National University Illustrated Pain Scale evaluated after 48 hours after surgery. Each item is scored using illustrations that corresponds to 0-10 levels of traumatic pain, beginning from 'no injury and/or pain' to 'causalgia'.
Postoperative Consumption of Patient-Controlled and/or Rescue Analgesics | 24 hours after surgery
  Amount of analgesics consumed through intravenous patient-controlled analgesia and/or administration of rescue analgesics
Postoperative Consumption of Patient-Controlled and/or Rescue Analgesics | 24.5 hours after surgery
  Amount of analgesics consumed through intravenous patient-controlled analgesia and/or administration of rescue analgesics
Postoperative Consumption of Patient-Controlled and/or Rescue Analgesics | 48 hours after surgery
  Amount of analgesics consumed through intravenous patient-controlled analgesia and/or administration of rescue analgesics
Understandability of Pain Scales | 48 hours after surgery
  Survey among patients on understandability pain scales
Convenience of Pain Scales | 48 hours after surgery
  Survey among patients on convenience of pain scales
Patient Satisfaction of Postoperative Pain Management | 48 hours after surgery
  Survey among patients on their level of overall satisfaction on postoperative pain management

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Jensen MP, Karoly P, Braver S. The measurement of clinical pain intensity: a comparison of six methods. Pain. 1986 Oct;27(1):117-126. doi: 10.1016/0304-3959(86)90228-9. PMID 3785962
- [Background] Breivik H, Borchgrevink PC, Allen SM, Rosseland LA, Romundstad L, Hals EK, Kvarstein G, Stubhaug A. Assessment of pain. Br J Anaesth. 2008 Jul;101(1):17-24. doi: 10.1093/bja/aen103. Epub 2008 May 16. PMID 18487245
- [Background] Karcioglu O, Topacoglu H, Dikme O, Dikme O. A systematic review of the pain scales in adults: Which to use? Am J Emerg Med. 2018 Apr;36(4):707-714. doi: 10.1016/j.ajem.2018.01.008. Epub 2018 Jan 6. PMID 29321111
- [Background] Pathak A, Sharma S, Jensen MP. The utility and validity of pain intensity rating scales for use in developing countries. Pain Rep. 2018 Aug 6;3(5):e672. doi: 10.1097/PR9.0000000000000672. eCollection 2018 Sep-Oct. PMID 30534623
- [Background] Eriksson K, Wikstrom L, Arestedt K, Fridlund B, Brostrom A. Numeric rating scale: patients' perceptions of its use in postoperative pain assessments. Appl Nurs Res. 2014 Feb;27(1):41-6. doi: 10.1016/j.apnr.2013.10.006. Epub 2013 Oct 31. PMID 24332467
- [Background] Noble B, Clark D, Meldrum M, ten Have H, Seymour J, Winslow M, Paz S. The measurement of pain, 1945-2000. J Pain Symptom Manage. 2005 Jan;29(1):14-21. doi: 10.1016/j.jpainsymman.2004.08.007. PMID 15652435
- [Background] Bond MR, Pilowsky I. Subjective assessment of pain and its relationship to the administration of analgesics in patients with advanced cancer. J Psychosom Res. 1966 Sep;10(2):203-8. doi: 10.1016/0022-3999(66)90064-x. No abstract available. PMID 4165548
- [Background] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420
- [Background] Bodian CA, Freedman G, Hossain S, Eisenkraft JB, Beilin Y. The visual analog scale for pain: clinical significance in postoperative patients. Anesthesiology. 2001 Dec;95(6):1356-61. doi: 10.1097/00000542-200112000-00013. PMID 11748392
- [Background] Katz J, Melzack R. Measurement of pain. Surg Clin North Am. 1999 Apr;79(2):231-52. doi: 10.1016/s0039-6109(05)70381-9. PMID 10352653
- [Background] Singer T, Seymour B, O'Doherty J, Kaube H, Dolan RJ, Frith CD. Empathy for pain involves the affective but not sensory components of pain. Science. 2004 Feb 20;303(5661):1157-62. doi: 10.1126/science.1093535. PMID 14976305